CLINICAL TRIAL: NCT03861286
Title: Characterisation of the Haemostatic Changes In Patients Receiving Intravenous Heparin for Cardiopulmonary Bypass Surgery
Brief Title: Haemostatic Markers in Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, deepa Jayakody Arachchillage, Consultant Haematologist, Imperial College London
Other Study IDs: 248558
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Unfractionated Heparin; Cardiopulmonary Bypass Surgery
Keywords: Cardiopulmonary Bypass Surgery; Unfractionated Heparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to understand the changes occurring in a blood clotting protein, von Willebrand factor (VWF), in patients undergoing cardiac surgery who receive the blood thinner called Heparin. These patients are given Heparin through their veins, to prevent blood clot formation as it passes through the heart bypass machine. At the end of the operation, the effect of Heparin is reversed by another drug, Protamine Sulphate.

Heparin prevents blood clots forming mainly by inactivating thrombin, a crucial protein needed for blood clotting. This effect of Heparin is monitored through blood tests called the 'Anti Factor-Xa' and the 'APTT'.

Heparin has another effect on clotting: it can block the attachment of special blood cell fragments called platelets to damaged blood vessels, but this effect is not usually measured.

Following blood vessel injury, the large VWF sticks to the damaged surface and captures platelets to form a 'plug' which stops bleeding. The platelet plug is then stabilised by other clotting proteins. This stops blood loss and allows vessel repair underneath.

Heparin blocks the ability of VWF to capture platelets at the site of blood vessel injury. The higher the dose of Heparin, the greater this blocking effect is. This secondary effect of Heparin cannot be readily monitored and may explain why bleeding complications occur in patients receiving Heparin despite the monitoring with blood tests used.

This study will look at the blood levels of Heparin, VWF and platelets before, during and after surgery and how well VWF functions in the presence of heparin, including its ability to attach to platelets.

The investigators will determine if all of the heparin related changes in blood clotting can be detected using a method that looks at all of the different steps in forming a blood clot.

DETAILED DESCRIPTION:
Von Willebrand factor (VWF) is a large plasma glycoprotein involved in thrombosis, haemostasis and vascular biology. Its principal role is to capture platelets at sites of blood vessel endothelial injury allowing the formation of an unstable platelet plug, an initial step in haemorrhage control. Following this, blood coagulation at the site of injury, results in the formation of fibrin strands, which enmesh and stabilise the platelet plug, until vessel repair is complete.

Following endothelial cell (EC) injury or activation, VWF becomes tethered, either to EC or to the now exposed subendothelial matrix (SEM). The shear stress generated by blood flow causes the tethered VWF to unravel, exposing its multiple platelet binding sites, resulting in platelet capture.

One of the most important domains of VWF is the A1 domain, which contains binding sites for the platelet receptor glycoprotein Ib (GPIb) as well as for collagen and heparin.

Heparin is the major component of mast cell secretory granules. Its precise physiological role is unknown but it has been proposed that it plays a role in host defense mechanisms. The anticoagulant properties of heparin, however, have been exploited pharmaceutically and exogenous heparin has been a clinically useful anticoagulant since 1935.4 It is known to potentiate the effects of antithrombin in the inactivation of Factor Xa and thrombin. Unfractionated heparin therapy can be monitored using the plasma activated partial thromboplastin time (APTT), anti -factor Xa activity or, if very high doses are used, the activated clotting time (ACT). The APTT is most commonly used to monitor UFH therapy as it is cost effective and readily available. However, it is subject to several pre-analytical and analytical variables and therefore may not provide an accurate measure of the anticoagulant effect of UFH. The anti-factor Xa activity is less susceptible to confounding factors and makes this the assay of choice but it is less widely available.

Studies have shown that heparin also competitively inhibits the binding of VWF to platelet receptor GPIb, an anti-thrombotic effect distinct from its anticoagulant role via Antithrombin. This may in part explain why the bleeding complications that occur during heparin therapy are unpredictable, despite using current techniques for monitoring its anticoagulant effect. This additional activity of heparin is likely to be of particular importance during CPB when very high concentrations of heparin are used to maintain the extracorporeal circuit and which have to be reversed to restore haemostasis at the end of the procedure. The currently available literature remains incomplete in the characterisation of the changes that occur in VWF-dependent platelet function and do not explain the observed recovery of VWF function above baseline levels, after reversal of heparin with protamine sulphate. The aim of this study is to fully characterise the changes in VWF concentration, function and platelet interaction, that occur in patients undergoing cardiac surgery and receiving intravenous unfractionated heparin, intra- and post-operatively. This is a prospective, single centre cohort study involving the analysis of haemostatic assays in patients receiving IV heparin during cardiopulmonary bypass surgery. The study aims to recruit 30 eligible adult patients (>18 years) undergoing first time cardiac surgery for the correction of atrial septal defects or undergoing tissue mitral valve replacement and receiving IV unfractionated heparin intra-operatively at Royal Brompton Hospital. The study aims to recruit a uniform population of 30 patients which should be achieved within 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing first time cardiopulmonary bypass surgery for correction of atrial septal defects or tissue mitral valve repair
2. Receiving intravenous Heparin for cardiopulmonary bypass

Exclusion Criteria:

* Concomitant Aortic Stenosis which is associated with an acquired von Willebrand Syndrome (aVWS)
* Patients with a baseline platelet count of <100x109/L
* Patients with a known coagulation factor deficiency or platelet function disorder
* Patients receiving heparin therapy prior to CPB within last 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort study, and patients undergoing cardiopulmonary bypass surgery will be recruited when they are assessed pre operatively at the Royal Brompton Hospital (RBH) Normal controls will be staff members from Imperial College London.
  Patient recruitment:
  Patients who meet the inclusion criteria will be identified by the anaesthetic team when they are assessed preoperatively. They will be provided with a Participant Information Sheet and have the opportunity to ask questions and discuss the study with the researchers before providing consent. The study aims to recruit 30 patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Quantitative & Qualitative VWF Assessment | 6 months
  VWF antigen level, Ristocetin Cofactor Assay

SECONDARY OUTCOMES:
Global Test of Haemostasis | 6 months
  Thromboelastography

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Arachachillage, MBBS, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sobel M, McNeill PM, Carlson PL, Kermode JC, Adelman B, Conroy R, Marques D. Heparin inhibition of von Willebrand factor-dependent platelet function in vitro and in vivo. J Clin Invest. 1991 May;87(5):1787-93. doi: 10.1172/JCI115198. PMID 2022745